CLINICAL TRIAL: NCT00267709
Title: A Phase 2a, Open-label Study of Visilizumab for Treatment of Perianal Fistulas in Patients With Crohn's Disease
Brief Title: Visilizumab for Treatment of Perianal Fistulas in Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Collaborators: PDL BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 291-411
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — visilizumab

INTERVENTIONS:
Drug: Visilizumab

SUMMARY:
The purpose of the study is to evaluate an intravenous (by injection) investigational medication to treat Crohn's disease in patients with at least one perianal fistula. The research is being conducted at up to 5 clinical research sites in the US and Europe and is open to both men and women ages 18 to 70 years old. Participants in the study will have a number of visits to a research site over a 17 month period. All study-related care and medication is provided to qualified participants at no cost: this includes all visits, examinations and laboratory work.

Visilizumab is a humanized antibody (antibodies are proteins that are normally made by the immune system to help defend the body from infections and other foreign substances) that is directed against T cells. Visilizumab selectively attacks problematic T cells and, in doing so, it may prevent them from causing inflammation. Visilizumab has also been observed to have a suppressive effect on the body's immune system (system in the body that reacts to foreign or occasionally one's own proteins).

DETAILED DESCRIPTION:
PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Diagnosis of Crohn's disease with fistula
* Test negative for Clostridium difficile within 3 weeks
* Signed informed consent, including permission to use protected health information.

Exclusion Criteria:

* History of lymphoproliferative disorder or prior malignancy within 5 years or current malignancy
* Pregnant or nursing
* HIV, Hepatitis B or Hepatitis C infection
* Presence of obstructive symptoms, confirmed by endoscopy, within 6 months
* Likely to require surgery in the next 6 months
* Serious or active infections within 1 year
* Active infections that require antibiotic therapy
* Serious infections that require IV antibiotics or hospitalization within 8 weeks
* Started or changed dose of sulfasalazine, 5-aminosalicylic acid (5-ASA), antibiotics, probiotics, or topical therapies for Crohn's within 2 weeks
* Had increased dose of corticosteroids within 2 weeks
* Received a live vaccine within 6 weeks
* Received any monoclonal antibodies or investigational agents within 3 months
* Received cyclosporine or tacrolimus (FK506) within 4 weeks
* Dose change or discontinuation of 6-mercaptopurine, azathioprine, or methotrexate within 4 weeks
* Significant organ dysfunction
* History of lymphoproliferative disorder
* History of tuberculosis, mycobacterial infection, or positive chest x-ray
* History of thrombophlebitis or pulmonary embolus
* History of immune deficiency or autoimmune disorders (other than Crohn's disease)
* History of seizure with subtherapeutic levels of anticonvulsive medication within one week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Clinical response, defined as external closure of at least 50% of perianal fistulas, without an accompanying increase in dose of concomitant medications, the addition of new medications, or Crohn's Disease-related surgery.

SECONDARY OUTCOMES:
Frequency of complete clinical response, confirm internal healing by MRI, duration of disease improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States